CLINICAL TRIAL: NCT01008345
Title: Effect of Ezetimibe on Oxidized LDL Cholesterol
Brief Title: Effect of Ezetimibe on Oxidized Low-density Lipoprotein (LDL) Cholesterol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hotel Dieu de France Hospital (Other)
Collaborators: Pharmaline, Lebanon (Unknown)
Responsible Party: Rabih Azar, MD, Hotel Dieu de France Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: pharmaline1
Record Dates: First submitted 2009-11-04; First posted 2009-11-05 (Estimated); Last update posted 2009-11-06 (Estimated); Status verified 2009-11

CONDITIONS: Coronary Artery Disease; Diabetes
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ezetimibe (Experimental): will receive the active treatment with ezetimibe and statin
  Interventions: Drug: ezetimibe
- placebo (Placebo Comparator)
  Interventions: Drug: ezetimibe

INTERVENTIONS:
Drug: ezetimibe — Patients will receive 10 mg/day of ezetimibe for 8 weeks

SUMMARY:
Randomized study. Patients with coronary artery disease equivalent will be randomized to receive atorvastatin 40 mg/day + placebo vs. atorvastatin 40 mg/day + ezetimibe 40 mg/day. Oxidized LDL cholesterol will be measured at baseline and after 8 weeks of treatment. Hypothesis is that ezetimibe will lower oxidized LDL

ELIGIBILITY:
Inclusion Criteria:

* CAD or CAD equivalent

Exclusion Criteria:

* Prior CABG or PCI within 3 months Prior use of ezetimibe within 3 months Receiving atorvastatin 40 mg/day or 80 mg/day or any dose of rosuvastatin CHF NYHA stage >2 Creatinin clearance < 30 ml/min

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
level of oxidized LDL cholesterol at end of study | 8 weeks of treatment

SECONDARY OUTCOMES:
small dense LDL level | 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: rabih azar, md, Principal Investigator — Hotel Dieu
Locations (1):
- Hotel Dieu de France Hospital, El Achrafiyé, Beyrouth, Lebanon